CLINICAL TRIAL: NCT03314779
Title: Continuous Monitoring of Cerebral Metabolic State. Combined Intracerebral and Jugular Bulb Microdialysis in Neurocritical Care.
Brief Title: Combined Intracerebral and Jugular Bulb Microdialysis
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Collaborators: Region of Southern Denmark (Other)
Responsible Party: Principal Investigator, Axel Forsse, MD, PhD-fellow, Odense University Hospital
Other Study IDs: 20150173
Record Dates: First submitted 2017-09-12; First posted 2017-10-19 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Subarachnoid Hemorrhage; Hypoxia Ischemia, Cerebral; TBI; Meningitis
MeSH Terms: conditions — Subarachnoid Hemorrhage; Hypoxia-Ischemia, Brain; Meningitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The first aim of this study is to investigate the frequency and severity of a specific pathological metabolic pattern, mitochondrial dysfunction, of the brain in comatose patients under neurocritical care. This pattern is recognized as a complication after compromised blood flow to the brain and may be amenable to treatment. The other main aim of this study is to correlate patterns of metabolites between brain and jugular venous blood. It is probable but not proven that jugular venous microdialysis can mirror the global metabolic state of the brain.

DETAILED DESCRIPTION:
Purpose

To describe the incidence of cerebral mitochondrial dysfunction in comatose patients admitted to the Neurointensive Care Unit (NICU) at Odense University Hospital and to evaluate the possible correlations between cerebral and jugular bulb microdialysis in an effort to develop new, effective and less invasive diagnostical tools for relevant patient groups.

Background

The hallmark of several serious neurological and neurosurgical disorders including severe traumatic brain injury, intracranial haemorrhage, cerebral infection and global hypoxic injury after cardiac arrest, is that the primary insult is out of reach for therapeutic intervention. Secondary injuries however, ensuing in the days to weeks after the primary insult are amenable to prevention or treatment. Inflammation, transient ischemia, free radical formation, cellular Ca2+-influx and mitochondrial dysfunction are therefore all examples of current research topics in neurointensive care.

The research group has a long history of experimental and clinical work in the area of cerebral metabolism in neurocritical disease. In recent years neuromonitoring with cerebral microdialysis has been a main focus, as well as mitochondrial dysfunction as a possible therapeutic target . In 2004 the investigators showed how monitoring SAH-patients with cerebral microdialysis could predict delayed neurological deterioration/vasospasm related complications, results that were corroborated by later external studies. In 2012 and 2014, results have been published showing how to diagnose mitochondrial dysfunction on the basis of the biochemical patterns of cerebral microdialysis experimentally as well as clinically. Briefly, a cerebrochemical pattern with elevated lactate/pyruvate-ratio with simultaneous normal or supranormal levels of pyruvate and glucose seen together with normal tissue oxygen monitoring indicates mitochondrial dysfunction. Mitochondrial dysfunction most likely plays a key role in the worsening of outcome in a variety cerebral pathological conditions, and might be amenable to pharmacologic intervention.

The microdialysis technique is based on a thin probe with a semipermeable membrane being inserted in affected brain tissue, collecting interstitial fluid from a small area surrounding the probe. The fluid is analysed for metabolites, proteins or pharmacological substances and has earlier been shown to be of great value in guiding NICU care and prognostication. One problem with the technique is, however, that the measurements are regional and limited to the very small sampling volume of the probe. Another obstacle is that the technique is intracranial invasive.

Aims

In the current prospective cohort study, the investigators will describe the incidence of mitochondrial dysfunction in a patients admitted to the NICU with severe subarachnoid haemorrhage (SAH). As patients suffering from SAH often have a non-ischemic cerebral metabolic affliction, a global cerebral measurement would presumably be as useful or more so than a focal measurement from only a very small regional brain volume. The investigators wish to evaluate a new method of monitoring, namely microdialysis of cerebral venous blood drainage. The cerebral venous drainage passes almost without exception through the jugular bulbs, left or right sided majority depending on dominance. The investigators will compare results of regional cerebral and venous measurements in order to confirm the hypothesis that metabolic disturbances of the brain are mirrored in the venous blood drainage in the jugular bulb. A pilot study of patients undergoing open heart surgery has confirmed significant differences in lactate and pyruvate in arterial systemic vs jugular venous blood. Yet unpublished data from this groups porcine experimental model supports the possibility of global metabolic venous monitoring.

Perspectives

If jugular bulb microdialysis can be confirmed to give a reliable global estimate of cerebral metabolic state it might be possible to a implement a new, less invasive diagnostic tool for NICU-patients. Surrogate measures in use today as e.g. NIRS (Near Infrared Spectroscopy) correlate poorly to cerebral metabolic status.

ELIGIBILITY:
Inclusion Criteria:

* Glasgow coma score <8.
* Suspicion of intracranial pathology

Exclusion Criteria:

* Suspected and/or Untreated coagulopathy
* Consent from closest of kin not given

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the neurointensive care unit at Odense University Hospital.
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2017-08-28 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Correlations of lactate/pyruvate-ratio (LP-ratio) calculated by dividing lactate concentration in mM by pyruvate concentration in mikroM, in cerebral and venous microdialysis | Patients are monitored a mean of 5 days with hourly analysis.
  Hourly samples of lactate (mM) and pyruvate (mikroM) are assessed using microdialysis measurements in brain and jugular bulb. The LP-ratio is calculated and compared at each timepoint.

SECONDARY OUTCOMES:
Correlations of microdialysis values of glucose. | Mean 5 day measurements
  Cerebral and jugular bulb microdialysis measurements of glucose (mM)compared for co-variation.
Modified Rankin scale of outcome. | 6 months
  6 month modified Rankin Scale (mRS) will be assessed at outpatient clinic. The mRS is the most widely used scale for measuring degree of disability in stroke trials, The scale ranges from 0 to 6, where 0 means no symptoms and 6 is dead.
Evaluation of mitochondrial dysfunction under study period. | calculations based on mean 5-day measurements per patient.
  Microdialysis results will be analysed for amount (hours) of mitochondrial dysfunction, defined as normal cerebral P02-measurements (mmHg), in combination with high LP-ratio (ratio) and simultaneous normal or high pyruvate concentration (mikroM).

CONTACTS AND LOCATIONS:
Overall Officials: Frantz Rom Poulsen, MD, PhD, Study Chair — Consultant, Professor, Research leader
Locations (1):
- Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nordstrom CH, Koskinen LO, Olivecrona M. Aspects on the Physiological and Biochemical Foundations of Neurocritical Care. Front Neurol. 2017 Jun 19;8:274. doi: 10.3389/fneur.2017.00274. eCollection 2017. PMID 28674514
- [Background] Nordstrom CH, Rehncrona S, Siesjo BK. Restitution of cerebral energy state, as well as of glycolytic metabolites, citric acid cycle intermediates and associated amino acids after 30 minutes of complete ischemia in rats anaesthetized with nitrous oxide or phenobarbital. J Neurochem. 1978 Feb;30(2):479-86. doi: 10.1111/j.1471-4159.1978.tb06553.x. No abstract available. PMID 624953
- [Background] Jacobsen A, Nielsen TH, Nilsson O, Schalen W, Nordstrom CH. Bedside diagnosis of mitochondrial dysfunction in aneurysmal subarachnoid hemorrhage. Acta Neurol Scand. 2014 Sep;130(3):156-63. doi: 10.1111/ane.12258. Epub 2014 May 3. PMID 24796605
- [Background] Nielsen TH, Olsen NV, Toft P, Nordstrom CH. Cerebral energy metabolism during mitochondrial dysfunction induced by cyanide in piglets. Acta Anaesthesiol Scand. 2013 Jul;57(6):793-801. doi: 10.1111/aas.12092. Epub 2013 Mar 18. PMID 23495747
- [Background] Nielsen TH, Bindslev TT, Pedersen SM, Toft P, Olsen NV, Nordstrom CH. Cerebral energy metabolism during induced mitochondrial dysfunction. Acta Anaesthesiol Scand. 2013 Feb;57(2):229-35. doi: 10.1111/j.1399-6576.2012.02783.x. Epub 2012 Sep 28. PMID 23017022
- [Background] Poulsen FR, Schulz M, Jacobsen A, Andersen AB, Larsen L, Schalen W, Nielsen TH, Nordstrom CH. Bedside evaluation of cerebral energy metabolism in severe community-acquired bacterial meningitis. Neurocrit Care. 2015 Apr;22(2):221-8. doi: 10.1007/s12028-014-0057-x. PMID 25142826
- [Background] Skjoth-Rasmussen J, Schulz M, Kristensen SR, Bjerre P. Delayed neurological deficits detected by an ischemic pattern in the extracellular cerebral metabolites in patients with aneurysmal subarachnoid hemorrhage. J Neurosurg. 2004 Jan;100(1):8-15. doi: 10.3171/jns.2004.100.1.0008. PMID 14743906
- [Background] Rostami E, Engquist H, Howells T, Johnson U, Ronne-Engstrom E, Nilsson P, Hillered L, Lewen A, Enblad P. Early low cerebral blood flow and high cerebral lactate: prediction of delayed cerebral ischemia in subarachnoid hemorrhage. J Neurosurg. 2018 Jun;128(6):1762-1770. doi: 10.3171/2016.11.JNS161140. Epub 2017 Jun 2. PMID 28574309
- [Background] Hutchinson PJ, Jalloh I, Helmy A, Carpenter KL, Rostami E, Bellander BM, Boutelle MG, Chen JW, Claassen J, Dahyot-Fizelier C, Enblad P, Gallagher CN, Helbok R, Hillered L, Le Roux PD, Magnoni S, Mangat HS, Menon DK, Nordstrom CH, O'Phelan KH, Oddo M, Perez Barcena J, Robertson C, Ronne-Engstrom E, Sahuquillo J, Smith M, Stocchetti N, Belli A, Carpenter TA, Coles JP, Czosnyka M, Dizdar N, Goodman JC, Gupta AK, Nielsen TH, Marklund N, Montcriol A, O'Connell MT, Poca MA, Sarrafzadeh A, Shannon RJ, Skjoth-Rasmussen J, Smielewski P, Stover JF, Timofeev I, Vespa P, Zavala E, Ungerstedt U. Consensus statement from the 2014 International Microdialysis Forum. Intensive Care Med. 2015 Sep;41(9):1517-28. doi: 10.1007/s00134-015-3930-y. PMID 26194024
- [Background] Tachtsidis I, Tisdall MM, Pritchard C, Leung TS, Ghosh A, Elwell CE, Smith M. Analysis of the changes in the oxidation of brain tissue cytochrome-c-oxidase in traumatic brain injury patients during hypercapnoea: a broadband NIRS study. Adv Exp Med Biol. 2011;701:9-14. doi: 10.1007/978-1-4419-7756-4_2. PMID 21445763